CLINICAL TRIAL: NCT00725114
Title: A Multicentre , Randomized, Double-blind, Placebo-controlled, Parallel-design Trial of the Efficacy and Safety of Subcutaneous Tetrodotoxin (TTX) for Moderate to Severe Inadequately Controlled Cancer-related Pain
Brief Title: Safety & Efficacy Study of Subcutaneous Tetrodotoxin for Moderate to Severe Inadequately Controlled Cancer-related Pain
Acronym: TEC-006
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wex Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEC-006
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2012-08

CONDITIONS: Pain; Cancer
Keywords: due; cancer; treatment
MeSH Terms: conditions — Pain; Neoplasms | interventions — Tetrodotoxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tetrodotoxin (Active Comparator)
  Interventions: Biological: Tetrodotoxin
- Sugar injection (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Tetrodotoxin — 30 µg twice daily for 4 days
  Other Names: TTX
  Arms: Tetrodotoxin
Biological: Placebo — 2 mL subcutaneous injection twice daily for 4 days
  Arms: Sugar injection

SUMMARY:
Different pathophysiologic mechanisms are responsible for the development of chronic pain disorders. Pain pathways are triggered in part by ectopic discharges of voltage-sensitive sodium channels, which are in abundance in both the peripheral and the central nervous systems. Tetrodotoxin (TTX) is a selective blocker of Na+ channels and causes analgesia either by decreasing the propagation of action potentials by Na+ channels and/or by blocking of ectopic discharges associated with chronic pain. TTX is extracted from the puffer fish (fugu). Results from animal pharmacology studies revealed that TTX is a more potent analgesic than standard analgesic agents such as aspirin, morphine or meperidine.

At present, the management of severe cancer pain generally includes the use of opiates. This can often result in undesirable side effects, and treatment with this type of medication is not always effective. Because currently available pain-relieving therapy is unsatisfactory for many patients, there is a need for new therapeutic approaches for the management of moderate or severe cancer pain.

Recent studies indicate that intramuscular (into a muscle) or subcutaneous (under the skin) injections of tetrodotoxin (TTX) may reduce pain in cancer patients who did not respond to standard therapies.

The current proposed study (TEC-006) is designed to 1) demonstrate in a double-blind, placebo-controlled trial that the subcutaneous 30 μg b.i.d. dose of TTX for 4 days is effective in reducing pain outcome and improving quality of life; 2) characterize the onset and duration of analgesia, and 3) demonstrate that TTX is well tolerated in patients with inadequately controlled cancer-related pain.

DETAILED DESCRIPTION:
Study Objectives:

Male or female subjects with moderate to severe pain (related to cancer or cancer treatment)inadequately controlled by current therapy:

Primary Objectives:

* To compare the efficacy of subcutaneous tetrodotoxin treatment (TTX) with that of placebo as measured by:

  * pain outcome (pain intensity reduction or use of analgesics)
  * improvement in quality of life (physical and emotional functioning)
* To compare the safety of subcutaneous tetrodotoxin with that of placebo.

Secondary Objectives:

* To assess the onset of analgesic response of subcutaneous tetrodotoxin.
* To determine the duration of analgesic response associated with subcutaneous tetrodotoxin treatment.

Overall Study Design:

This will be a multicentre, randomized, double-blind, placebo-controlled, parallel-design trial of the efficacy and safety of tetrodotoxin in patients over 18 years of age with stable but inadequately controlled moderate to severe pain associated with cancer. Approximately 15 centers across Canada, New Zealand and Australia are expected to participate. Subcutaneous tetrodotoxin (30 µg b.i.d.) or placebo will be administered to 127 patients per group for four consecutive days.

The study period will be at least three weeks from the start of screening to the end of analgesic response. Patients will be screened for the study and will enter a 4- to 7-day baseline period within 28 days of screening. Following the baseline period, patients will either be admitted to the hospital or be seen at the site's outpatient facility on a daily basis. Patients will be randomized on Day 1 to receive study drug twice daily for four consecutive days. After the treatment period, all patients will be seen again on Days 5, 8, and 15 for further safety and efficacy evaluations, and then every two weeks until their pain returns.

Sample Size:

A total of 254 subjects (127 per treatment arm) will be enrolled in this study. The first interim analysis is planned to adjust the sample size after 60 evaluable subjects are enrolled, completed and data are available for analysis. A second interim analysis is planned after 50% of subjects(110 evaluable subjects) have completed the study and data are available for analysis.

Investigational Product 30 µg TTX (tetrodotoxin injectable) or an equivalent volume of placebo, identical in appearance, injected subcutaneously twice daily for 4 days.

Efficacy Variables:

Efficacy assessments will include global pain intensity, component-specific pain intensity, ATC and breakthrough analgesic use, impact of pain on physical functioning (general activity, walking ability, or normal work), and emotional functioning (mood, relations with other people, or enjoyment of life), impressions of change, onset of analgesic response, duration of analgesic response, and time to peak analgesic response.

Safety Variables:

Safety assessments will include adverse event reporting, vital signs, physical and neurological examinations, 12-lead electrocardiogram, clinical laboratory tests.

Data Analysis Method:

Two co-primary endpoints will be analyzed in this study as follows:

Co-primary #1 (composite endpoint): Proportion of responders observed in each treatment arm for the composite endpoint satisfying the following three components:

1. a ≥30% decrease in mean pain intensity or a decrease of ≥50% of opioid use from baseline
2. a ≥30% improvement of QOL in at least one descriptor of physical functioning
3. a ≥30% improvement of QOL in at least one descriptor of emotional functioning

Co-primary #2 (Pain intensity endpoint): Proportion of responders observed in each treatment arm for reduction in pain intensity satisfying the following:

1. a ≥30% decrease in mean pain intensity or a decrease of ≥50% of opioid use from baseline

Trends for differences between treatments will be individually tabulated for:

* impact of pain on physical functioning
* impact of pain on emotional functioning

Comparison of the proportion of responders in each treatment group will be made using the Mantel-Haenszel procedure.

Safety as assessed by the analysis of adverse events, abnormal laboratory results, and abnormalities detected by 12-lead electrocardiogram.

ELIGIBILITY:
Inclusion criteria

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Male or female 18 years of age and over.
2. Inpatient or outpatient with a diagnosis of cancer.
3. Stable but inadequately controlled pain with current therapy for at least two weeks.
4. Experiencing somatic, visceral and/or neuropathic pain related to cancer.
5. Baseline pain intensity, as assessed by Question #3 of the Brief Pain Inventory (BPI) that meets the definition of "moderate" (score of 4-5) or "severe" (score of 6-10) pain.
6. Life expectancy of at least 3 months.
7. Ability to communicate well with the investigator and to comply with the requirements (restrictions, appointments, and examination schedule) of the entire study.
8. Signed informed consent document (prior to any study-related procedures being performed).

Exclusion criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Planned initiation of chemotherapy, radiotherapy, or bisphosphonates within 30 days prior to randomization.
2. Use of anaesthetics.
3. Use of lidocaine and other types of antiarrhythmic drugs.
4. Use of scopolamine and acetylcholinesterase-inhibiting drugs such as physostigmine.
5. History of CO2 retention, or SaO2 <80% either on room air or O2 of not greater than 2-4 L/min by nasal cannula.
6. Second- or third-degree heart block or prolonged QTc interval (corrected for rate) on screening ECG (confirmed > 450 msec on repeated occasion) or any other active cardiac arrhythmia or abnormality that could constitute a clinical risk.
7. Coagulation or bleeding defects if, in the opinion of the investigator, this represents a risk to the subject considering the subcutaneous (s.c.) route of administration.
8. Known hypersensitivity to puffer fish, tetrodotoxin and/or its derivatives.
9. Use of an investigational agent within 30 days prior to screening or is scheduled to receive an investigational drug other than tetrodotoxin during the course of the study.
10. Females who are lactating or at risk of pregnancy (i.e., sexually active with fertile males and not using an adequate form of birth control).
11. Females with a positive serum pregnancy test at screening or positive urine pregnancy test on admission to study site.
12. Any other condition that, in the opinion of the investigators, is likely to interfere with the successful collection of the measures required for the study or poses a risk to the patient.
13. Men with glomerular filtration rate (GRF) less than 60 mL/min/1.73 m2 and women with GFR less than 50 mL/min/1.73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2008-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Efficacy: Composite-endpoint will be an evaluation that combines pain outcome and quality of life. Pain intensity will be used a co-primary endpoint. Safety as assessed by the analysis of AEs, 12-lead ECG, and abnormal lab values. | Dec2010

SECONDARY OUTCOMES:
The period of onset of pain response as reported by responders. | Dec2010
The number of days a subject meets the definition of pain response. | Dec2010

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Neil Hagen, MD, FRCPC, Study Chair — Tom Baker Cancer Centre
Locations (1):
- WEX Pharmaceuticals Inc., Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Hagen NA, Cantin L, Constant J, Haller T, Blaise G, Ong-Lam M, du Souich P, Korz W, Lapointe B. Tetrodotoxin for Moderate to Severe Cancer-Related Pain: A Multicentre, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design Trial. Pain Res Manag. 2017;2017:7212713. doi: 10.1155/2017/7212713. Epub 2017 May 7. PMID 28555092